CLINICAL TRIAL: NCT06907303
Title: Development and Evaluation of RNA-based Markers for Detecting and Diagnosing Endometriosis
Brief Title: RNA Assays for Endometriosis Detection and Diagnosis
Acronym: RNA-EndoDx
Status: Enrolling by invitation | Type: Observational
Sponsor: Wren Laboratories LLC (Industry)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Other Study IDs: WrenEndoMstudy 01
Record Dates: First submitted 2025-03-25; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis
Keywords: Endometriosis; Diagnosis; Gene Expression; PCR
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis: Women with suspected endometriosis undergoing laparoscopy to provide tissue for pathological diagnosis of the disease.
  Interventions: Diagnostic Test: EndoDx
- Control: Women undergoing surgery for benign cervical disease.
  Interventions: Diagnostic Test: EndoDx

INTERVENTIONS:
Diagnostic Test: EndoDx — PCR assay for Endometriosis diagnosis

SUMMARY:
Endometriosis is a common disease that affects up to 10% of women of reproductive age. Diagnosis, however, is typically delayed (up to 12 years) and is usually made after surgery. A key unmet need therefore is an accurate biomarker that can be used to detect the disease early. This study is a prospective trial to identify candidate mRNA-markers which can be used to aid in the diagnosis of this disease. It is a discovery/validation study that will identify and confirm a gene expression panel that is specific for endometriosis and provides a non-invasive tool for future use.

DETAILED DESCRIPTION:
Endometriosis is a common disease that affects up to 10% of women of reproductive age. Diagnosis, however, is typically delayed (up to 12 years) and is typically made after surgery. A key unmet need therefore is an accurate, non-invasive biomarker that can be used to detect the disease early.

We hypothesize that endometriosis-related circulating gene expression can be identified using transcriptomic and bioinformatics approaches and used to construct an accurate diagnostic tool for this condition.

The primary objective is to develop a gene signature that detects endometriosis. The hypothesis is that this disease is characterized by a set of genes that characterize endometriosis tumor biology.

The aim is to detect over-expressed genes (elevated mRNA expression) in endometriosis tissue. The goal is to identify 10-25 biomarker genes that are highly expressed to form a candidate biomarker panel.

Highly expressed genes will be determined against samples collected from age/menstrual stage matched controls. A bio-informatics approach will be used to identify these over-expressed genes. This form the basis of a potential diagnostic panel.

Per PICOT criteria:

* The target patient population are women aged 20-35 years with a pathological diagnosis of endometriosis.
* The intervention is sample collection at the time of diagnosis (tissue, blood, saliva)
* The comparison group are normo-ovulatory subjects (age 20-25 years) undergoing surgery for benign cervical lesions.
* The outcome is a gene signature that is associated with endometriosis.
* The follow-up time is one year.

The secondary objective is to test the diagnostic utility of the 10-25 gene panel. This will be undertaken using the retrospectively collected samples.

* Each of the highly expressed genes will be measured and quantified using an RT-PCR approach.
* Genes that are statistically over-expressed in the endometriosis samples will be selected for a PCR panel.
* The expression of genes in the PCR panel will be scored.
* Low scores will be related to "control" and higher scores to "endometriosis".
* The scores will be formally evaluated as a diagnostic (area under the curve analysis, accuracy, sensitivity and specificity metrics).
* A specific comparison will be made between the endometriosis cohort and the control cohort.
* The metrics for a successful assay are:

  * Accuracy >80%
  * Sensitivity >90%
  * Specificity >85%
  * AUC >0.8

ELIGIBILITY:
Inclusion Criteria:

For the endometriosis cohort

* a history of infertility more than 1 year
* age 20-35 years
* normal liver and kidney function, without gynaecological and other systemic disease

Inclusion criteria for controls include normo-ovulatory history, aged between 20-35 years, who exhibit normal liver and kidney function, and do not have any systemic diseases including autoimmune disease.

-

Exclusion Criteria:

For the endometriosis cohort

* polycystic ovary syndrome, hyperprolactinemia
* severe cardiovascular system, liver, kidney, and hematopoietic system disease
* autoimmune disease
* uterine fibroids, endometritis, non-vegetative ovarian cysts, ovarian malignancies, and internal genital tuberculosis

Exclusion criteria for the controls includes gynaecological malignancies and genital tuberculosis.

-

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Women with high suspicion of endometriosis and women undergoing surgery for benign cervical disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop a gene signature that detects endometriosis | 12-18 months
  Gene expression levels in samples from endometriosis subjects and controls

SECONDARY OUTCOMES:
Assess the diagnostic utility of the gene signature to differentiate between endometriosis and controls | 6 months
  Algorithmic analysed normalized gene expression levels in samples from endometriosis subjects and controls

CONTACTS AND LOCATIONS:
Locations (2):
- Wren Laboratories, Branford, Connecticut, United States
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No